CLINICAL TRIAL: NCT04926012
Title: Descriptive and Risk Factors Analysis of All-cause Postoperative Death in Patients Undergoing Cardiovascular Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: National Center for Chronic and Noncommunicable Disease Control and Prevention, China CDC (Other); Henan Provincial People's Hospital (Other); Xiangya Hospital (Other); Shanxi Bethune Hospital (Other)
Responsible Party: Principal Investigator, Shanglong Yao, Clinical Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: PODSV1
Record Dates: First submitted 2021-06-09; First posted 2021-06-14 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Postoperative Death
Keywords: Postoperative death; Cardiovascular surgery; Prediction model

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators are aimed to develop and externally validate a prediction model of clinical risk factors that quantifies postoperative death after cardiac and vascular surgery.

The investigators identify all patients treated with cardiovascular surgery, between 2000 and 2020, within the Wuhan Union hospital and all collaborators. The surgical patient cohort will be matched with the National Death database to determine the patient's postoperative death data.

60% patients were randomly selected to the development cohort. Logistic regression analysis for prediction of postoperative death adjusted for different covariates. The model was externally validated in the remaining 40% patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients Undergoing Cardiovascular Surgery

Exclusion Criteria:

* Patients with incomplete electronic medical record information

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients Undergoing Cardiovascular Surgery
Sampling Method: Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2021-07-30 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative Death | The mortality within 5 years after the cardiovascular surgery

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - National Center for Chronic and Noncommunicable Disease Control and Prevention, Chinese Center for Disease Control and Prevention, Beijing, Beijing Municipality
  - Henan People's Hospital, Henan, China, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangya Hospital, Hunan, China, Changsha, Hunan
  - Shanxi Bethune hospital, Shanxi, China, Taiyuan, Shanxi